CLINICAL TRIAL: NCT00022932
Title: Phase II Multicenter Study of Iodine-131 Anti-B1 Antibody Consolidation For Patients With Diffuse Large B-Cell Non-Hodgkin's Lymphoma Following First-Line CHOP
Brief Title: Safety and Efficacy of Iodine-131 Anti-B1 Antibody for Intermediate Grade Non-Hodgkin's Lymphoma Following First Line CHOP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Corixa Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-99-032
Record Dates: First submitted 2001-08-16; First posted 2001-08-20 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-09

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Non-Hodgkin's Lymphoma; Radioimmunotherapy; Monoclonal Antibody; Corixa; Bexxar; Anti-B1 Antibody; Tositumomab; Iodine -131 Anti-B1 Antibody; Iodine I 131 Tositumomab
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — tositumomab I-131

INTERVENTIONS:
Drug: Iodine-131 Anti-B1 Antibody

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of using Iodine-131 Anti-B1 Antibody for the treatment of patients with large B-cell non-Hodgkin's lymphoma (NHL) who have achieved a response following 6-8 cycles of CHOP therapy.

DETAILED DESCRIPTION:
The primary endpoint is to determine the incidence of Grade IV hematologic toxicity following Iodine-131 Anti-B1 Antibody consolidation for patients with diffuse large B-cell NHL who achieved a response (PR, CRu, CR) following first-line CHOP chemotherapy. The secondary efficacy endpoints are to determine the complete response rate, duration of response, duration of complete response, progression-free survival, and time to treatment failure. The pharmacokinetic endpoint is to determine the total body residence time following the dosimetric dose. The secondary safety endpoints are to determine the incidence of adverse experiences, hematologic toxicity (e.g., nadir, time to nadir, and time to recovery), use of supportive care, percent of patients converting to human anti-murine antibody (HAMA) positivity, and survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed initial diagnosis of de novo diffuse large B-cell NHL according to the REAL classification. This includes the intermediate grade International Working Formulation subtypes of diffuse, mixed small cell and large cell; diffuse large cell; follicular large cell; mantle cell, and large cell immunoblastic.
* Patients must have had Ann Arbor, stage III or stage IV, or bulky Stage II disease at diagnosis.
* Patients must be less than or equal to 80 years of age with any IPI score.
* Patients must have less than an average of 25% of the intratrabecular marrow space involved by NHL in bilateral bone marrow biopsy specimens as assessed microscopically at study entry. A unilateral bone marrow biopsy demonstrating <10% involvement with NHL is also adequate. Verification of bone marrow status must be performed at the time of response evaluation following CHOP chemotherapy and within 56 days of study enrollment.
* Patients must have been treated with 6 or more cycles of first-line CHOP chemotherapy and have achieved a PR, CRu, or CR. Patients must have available computed tomography (CT) scans of the chest, abdomen, and pelvis, and a bone marrow biopsy that were performed within 56 days prior to the start of CHOP. In addition, they must have written documentation (i.e., copies of original medical notes and radiographic reports) describing the pre-CHOP staging evaluation, the number of cycles of CHOP administered, the dose of each agent, the start and stop dates of each cycle, and the post-CHOP response evaluation. The post-CHOP response evaluation must include a CT scan of the chest, abdomen, and pelvis (gallium scan is optional). For patients who have palpable cervical lymphadenopathy, a CT scan of the neck must be performed following CHOP chemotherapy. The CHOP chemotherapy should consist of standard doses of each agent, although dose-reduction is permitted. CHOP cycle delay is also permitted.
* The patient must be enrolled within 56 days of the first day of the last cycle of CHOP chemotherapy and within 35 days following response evaluation after CHOP chemotherapy.
* Patients must have evidence that their tumor tissue expresses the CD20 antigen.
* Patients must have a performance status of at least 60% on the Karnofsky Performance Scale and an anticipated survival of at least 3 months.
* Patients must have an ANC greater than or equal to 1500 cells/mm3 and a platelet count greater than or equal to 100,000 cells/mm3 within 14 days of study enrollment. These blood counts must be sustained without support of hematopoietic cytokines or transfusion of blood products.
* Patients must have adequate renal function (defined as serum creatinine <1.5 times the upper limit of normal) and hepatic function (defined as total bilirubin less than or equal to 2.0 times the upper limit of normal and AST <5 times the upper limit of normal) within 20 days of study enrollment.
* Patients of childbearing potential must undergo a negative serum pregnancy test within 14 days prior to study enrollment

Exclusion Criteria:

* Patients who have received prior chemotherapy other than first-line CHOP. Patients must not have been treated with radiation, or biological therapy prior to or after CHOP chemotherapy.
* Patients with active bilateral obstructive hydronephrosis.
* Patients with New York Heart Association class III or IV heart disease or other serious illness that would preclude evaluation.
* Patients with prior malignancy other than lymphoma, except for adequately treated skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for 5 years. Patients who have been disease-free of another cancer for greater than 5 years must be carefully assessed at the time of study enrollment to rule out recurrent disease.
* Patients with known HIV infection.
* Patients who are HAMA positive.
* Patients with known brain or leptomeningeal metastases at any time since diagnosis.
* Patients with active infection requiring IV anti-infectives at the time of study enrollment.
* Patients who are pregnant or breastfeeding. Males and females must agree to use a contraceptive method from enrollment to 6 months after receiving Iodine-131 Anti-B1 Antibody.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Rush Medical Center, Chicago, Illinois
  - Tufts New England Medical Center, Boston, Massachusetts
  - Cornell Medical Center, New York, New York